CLINICAL TRIAL: NCT07101809
Title: Evaluating the Safety and Effectiveness of Steerable Ureteroscopic Renal Evacuation (SURE) With the CVAC® System Compared to Standard Ureteroscopy With no Suction for the Treatment of Renal Stones: a Prospective, Randomized Trial
Brief Title: Trial of Ureteroscopy vs Steerable Continuous Flow Aspiration Technology
Acronym: TRUST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Calyxo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP00006
Record Dates: First submitted 2025-07-25; First posted 2025-08-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Urolithiasis; Stones, Kidney; Renal Stones; Kidney Stones
Keywords: ureteroscopy; CVAC; SURE
MeSH Terms: conditions — Urolithiasis; Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Ureteroscopy (URS) (Active Comparator): This is a treatment in which the urologist uses a laser to break a kidney stone into very small pieces and then places a tool called a stent to allows the remaining pieces to fall out.
  Interventions: Device: Standard Ureteroscopy (URS)
- Steerable Ureteroscopic Renal Evacuation (SURE) with CVAC System (Active Comparator): The CVAC Aspiration System is a sterile, single use, steerable ureteral catheter system with integrated vision, irrigation and aspiration for the treatment and removal of urinary stones (kidney stones, fragments, and dust).
  Interventions: Device: Steerable Ureteroscopic Renal Evacuation (SURE) using the CVAC System

INTERVENTIONS:
Device: Steerable Ureteroscopic Renal Evacuation (SURE) using the CVAC System — The CVAC Aspiration System is a sterile, single use, steerable ureteral catheter system with integrated vision, irrigation and aspiration for the treatment and removal of urinary stones (kidney stones, fragments, and dust).
  Other Names: CVAC
  Arms: Steerable Ureteroscopic Renal Evacuation (SURE) with CVAC System
Device: Standard Ureteroscopy (URS) — Arm Description: This is a treatment in which the urologist uses a laser to break a kidney stone into very small pieces and then places a tool called a stent to allows the remaining pieces to fall out.
  Arms: Standard Ureteroscopy (URS)

SUMMARY:
The goal of this clinical trial is to compare Steerable Ureteroscopic Renal Evacuation (SURE) using the CVAC System and standard ureteroscopy (URS) with laser lithotripsy for the treatment of urolithiasis. This is a prospective, randomized (1:1), multi-center study.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for ureteroscopy with laser lithotripsy
* Be willing and able to return for and respond to all study-related follow up procedures
* Have been informed of the nature of the study and has provided informed consent using the IRB approved informed consent (ICF)

Exclusion Criteria:

* Untreated urinary tract infection at the time of the index procedure
* Significant comorbidities
* Bladder, ureteral or kidney abnormalities
* Pregnant individuals
* Unable to meet the treatment and follow up protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Residual Stone Volume (RSV) | 30-Day